CLINICAL TRIAL: NCT02849119
Title: Comparison of Peri-operative Outcomes of Laparoscopic or Robotic Partial Nephrectomy for Small Renal Mass: Transperitoneal vs Retroperitoneal Approach
Brief Title: Transperitoneal vs Retroperitoneal Laparoscopic or Robotic Partial Nephrectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2015-03-068-002
Record Dates: First submitted 2016-06-28; First posted 2016-07-29 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2015-09

CONDITIONS: Renal Cell Carcinoma
Keywords: Robot; Laparoscopic; Partial nephrectomy; Transperitoneal; Retroperitoneal; Laparoscopic Surgery; Surgical Procedures, Robotic; Nephrectomy
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Laparoscopy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transperitoneal approach (Experimental): Laparoscopic or Robotic Partial Nephrectomy through transperitoneal approach
  Interventions: Procedure: Laparoscopic or robotic partial nephrectomy
- Retroperitoneal approach (Experimental): Laparoscopic or Robotic Partial Nephrectomy through retroperitoneal approach
  Interventions: Procedure: Laparoscopic or robotic partial nephrectomy

INTERVENTIONS:
Procedure: Laparoscopic or robotic partial nephrectomy — Laparoscopic or robotic partial nephrectomy of a small renal masses (T1a) through transperitoneal or retroperitoneal approach

SUMMARY:
Both laparoscopic partial nephrectomy (LPN) and robotic partial nephrectomy (RPN) can be performed through transperitoneal (TP) or retroperitoneal (RP) approach. RP approach is less utilized than TP approach because of technical difficulties when using rigid laparoscopic instruments in the small space of retroperitoneum cavity. However, with advanced surgical skills and thoughtful patient selection, RP approach may be associated with shorter operative time (OT), less estimated blood loss (EBL), shorter length of hospital stay (LOS) compared with TP approach.

Therefore, the investigators performed randomized control trial to compare the outcomes of the two approaches (TP-LPN or RPN vs RP-LPN or RPN).

DETAILED DESCRIPTION:
Partial nephrectomy is the standard treatment for small renal masses. The evolution of minimally invasive partial nephrectomy led to widespread utilization of laparoscopic (LPN) and robotic partial nephrectomy (RPN). Both LPN and RPN can be performed through transperitoneal (TP) or retroperitoneal (RP) approach. RP approach is less utilized than TP approach because of technical difficulties when using rigid laparoscopic instruments in the small space of retroperitoneum cavity. However, with advanced surgical skills and thoughtful patient selection, RP approach may be associated with shorter OT, less EBL, shorter LOS compared with TP approach.

Therefore, the investigators performed randomized control trial to compare the outcomes of the two approaches (TP-LPN or RPN vs RP-LPN or RPN).

The purpose of this study To compare the treatment outcomes of the transperitoneal and retroperitoneal approach during LPN or RPN in treatment of small renal masses.

Inclusion criteria During the study period, a small renal mass (less than 4cm, T1a stage) patients are going to underwent LPN or RPN.

Exclusion criteria

1. Patients who underwent radical nephrectomy
2. Patients with bilateral renal masses
3. Patients with a solitary kidney
4. Patients reject a written informed consent
5. Pregnancy

The number of target subjects More than 106 patients who meet the inclusion criteria

ELIGIBILITY:
Inclusion Criteria:

* Patients are going to undergo LPN or RPN with renal mass =<4cm

Exclusion Criteria:

* Bilateral renal masses Solitary kidney Previous underwent nephrectomy refuse to be enrolled the study pregnancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Operative time | Intraoperative
  Operative time of partial nephrectomy

SECONDARY OUTCOMES:
Warm ischemic time (minutes) | Intraoperative
  Vessel clamping time during partial nephrectomy
Number of participants with treatment-related adverse events as assessed by Clavien-Dindo classification | from date of surgery, to 1 year postoperatively
Change of differential glomerular filtration rate (dGFR) measured by renal scan | Preoperative dGFR and postoperative 1 year
Overall disease-free survival time (month) | from date of surgery, to 1 year postoperatively
  Disease free means no local recurrence, no metastasis.

CONTACTS AND LOCATIONS:
Overall Officials: Seongil Seo, MD, Study Chair — Urology department of Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No